CLINICAL TRIAL: NCT03314311
Title: Rehabilitative Strategies Following Oesophageal Cancer
Acronym: ReStOre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Principal Investigator, Prof Juliette Hussey, Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRA-POR-2014-535
Record Dates: First submitted 2015-05-18; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Esophageal Cancer
Keywords: Rehabilitation; Exercise; Nutrition Therapy; Patient Education as Topic
MeSH Terms: conditions — Esophageal Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation Programme (Experimental): 12 week multi-disciplinary intervention prescribing exercise, individual dietary counselling and education sessions.
  Interventions: Behavioral: Rehabilitation programme
- Control (No Intervention): Usual care control arm

INTERVENTIONS:
Behavioral: Rehabilitation programme — The RESTORE trial is a 12 week multi-disciplinary intervention involving exercise, nutrition advice and education sessions
  Arms: Rehabilitation Programme

SUMMARY:
The ReStOre trial is a multi-disciplinary intervention of exercise, diet and education for patients who have completed treatment for oesophageal cancer. The intervention aims to improve quality of life and functional performance following oesophageal cancer and assist patients to return to normal activity during the early survivorship phase. The 12-week intervention will involve structured exercise training, individual dietary advice and multi-disciplinary education sessions addressing a range of survivorship needs.

DETAILED DESCRIPTION:
The principal study proposed in this work will be composed of two phases. Phase I will consist of a longitudinal analysis, tracking the progression of cachexia and associated dysmetabolic state throughout treatment for oesophageal cancer (OC) and examining the impact of this decline on measures of physical functioning. A total of 88 newly-diagnosed OC patients will be recruited for Phase I. In Phase II, participants from Phase I will be re-assessed and if deemed suitable, will be enrolled onto a multidisciplinary team rehabilitation programme aimed at improving functional status. This rehabilitation programme will take the form of a randomised controlled trial (RCT) and will be based on the well-established cardiac rehabilitation programme model. It is anticipated that approximately 50% of participants enrolled onto Phase I will be suitable for progression to Phase II.

Outcomes The primary outcome across both Phase I and Phase II is functional capacity. Secondary outcomes including inflammatory status, energy metabolism and nutritional status will be measured as appropriate during the study. All outcomes are discussed in detail elsewhere.

Phase I: Longitudinal Study Examining the impact of progressive cachexia, dysmetabolism and cancer treatment on functional capacity in OC patients

Phase I will be designed as a longitudinal analysis, commencing at the time of diagnosis, tracking the progression of cachexia and associated dysmetabolic state, incorporating inflammatory profiles, energy metabolism (oxidative phosphorylation and glycolysis) and gut hormones, throughout treatment for OC and examining the impact of this decline on measures of physical functioning. Assessments will be completed at diagnosis (T0), cycle 2 chemotherapy (T1), cycle 3 chemotherapy (T2), pre-oesophagectomy (T3), post-oesophagectomy (T4), 4-weeks post-surgery (T5) and six months post-surgery (T6). All assessments will be completed during the same day as routine out-patient appointments thereby reducing the burden on participants. Furthermore, blood samples will be taken during routine clinical sampling and CT scans will be completed as part of routine medical care.

Phase II: Randomised Controlled Trial Can rehabilitation following curative treatment for OC optimise health-related functional outcomes?

Phase II will examine the effect of a 12-week rehabilitation programme, incorporating a walking intervention, individualised nutritional advice and education session, on functional status following curative treatment for OC. Following completion of Phase I and medical clearance to progress to Phase II, participants will be randomised 1:1 to either the intervention group or a control group. The control group will not receive the intervention however following completion of final assessments, participants will be offered an individual exercise and dietary session with the research physiotherapist and dietitian. During the intervention period, participants in the control group will continue to receive routine medical care.

The primary outcome for the multidisciplinary rehabilitation programme will be a change in functional capacity as measured by aerobic capacity. Secondary measures of functional capacity will include a stair climbing test, hand grip and physical activity. Body composition will also be measured by bio impedance analysis. The secondary outcomes that will be assessed are nutritional status, dietary quality and healthy related quality of life (QOL). Inflammatory profiles, measures of energy metabolism and gut hormones are unlikely to be influenced by the proposed rehabilitative intervention and therefore will not be measured. Assessments will be completed at, programme completion and three months post programme completion. Assessments take place at the Welcome Trust-HRB Clinical Research Facility St. James's Hospital. The rehabilitation programme will consist of three main components; 1. Exercise session, 2. Dietary sessions and 3. Education sessions. The intervention outlined below is devised based best evidence, pilot data and clinical expertise. The design final design will be informed form the results of the feasibility study and from needs identified in Phase I.

Exercise Sessions The exercise component of the rehabilitation programme will take the form of a 12 week supervised and home-based walking intervention. A walking intervention was chosen as walking is the most common form of exercise completed by adults nationally and worldwide, it is safe and feasible for deconditioned cohorts and represents a functionally meaningful activity. The feasibility of implementing a similar programme in cancer survivors has been previous established.

Group walking sessions will be supervised twice weekly during the first four weeks of the programme to re-introduce exercise to participant's lives in a safe and structured manner. As the programme progresses the frequency of supervised sessions will decrease to increase participants independence with the protocol. In the absence of guidance on appropriate exercise prescription in cancer cohorts, exercise intensity will be prescribed in accordance with the American College of Sports Medicine (ACSM) guidelines for exercise in deconditioned populations (28). Initially, activity will be prescribed at a light intensity and will progress during the programme to a moderate aerobic intensity. The proposed starting intensity is based on pilot data from the investigators institute suggesting that aerobic fitness levels are either 'poor' or 'very poor' in the early post-treatment phase. Participants will wear Polar Heart Rate monitors during all sessions to ensure compliance with the exercise prescribed. The goal at programme completion will be participation in 30 minutes of moderate intensity activity five days per week, as per the ACSM physical activity guidelines.

Nutrition Sessions Nutrition sessions will be delivered during week 1, week 2 and then fortnightly on a one to one basis. Weight and circumferential measures will be recorded at each session and dietary intake will be assessed as described previously.

The education delivered in the nutrition sessions will be individualised to participants needs. There is limited knowledge of the specific nutritional needs of oesophageal cancer survivors. Based on experience at this centre, the investigators anticipate that a heterogeneous mix of dietary issues requiring intervention will present in this cohort. These include persistent weight loss, anorexia, gastrointestinal disturbance and altered bowel habit. In addition, participants may require specific dietary advice to reduce the risk of other diseases e.g. cardio-protective dietary advice. Furthermore, the increase in physical activity by participants throughout the intervention will require dietary monitoring and advice to avoid inappropriate negative energy balance.

The feasibility study will assist in identifying specific nutritional issues facing oesophageal cancer survivors and help inform content and delivery of the nutrition education sessions. The target for participants is optimal dietary intake in line with the WCRF guidelines for cancer survivors. Supporting literature detailing prescriptive dietary advice will be developed and provided to participants.

Education Sessions Education sessions will be delivered weekly during weeks 1-4 and fortnightly thereafter by a range of members of the multidisciplinary team. As per the cardiac rehabilitation model, education sessions will talk place after the exercise session and cool-down, to monitor participant recovery following exercise. Education topics covered by the physiotherapist will include advice regarding physical activity guidelines, discouraging sedentary behaviour and overcoming barriers to physical activity. The dietitian will discuss dietary management of gastrointestinal symptoms and will also educate participants on healthy eating for cancer survivors as per World Cancer Research Fund, including practical advice and strategies to achieve dietary goals. Participants will be encouraged to highlight topics that may be of particular concern to them for discussion. As per the cardiac rehabilitation model, such topics may be covered by members of the multi-disciplinary team including the surgeon, gastrointestinal nurse, occupational therapist or social worker. Education sessions will take place at the Welcome Trust-HRB Clinical Research Facility St. James's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed treatment for oesophageal cancer to include oesophagectomy. Patients may have also been treated with neo-adjuvant or adjuvant chemotherapy or chemoradiotherapy.
* Curative treatment intent.
* Age >18 years
* Able to understand English

Exclusion Criteria:

* Evidence of active or recurrent disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in Aerobic Fitness | Change from baseline in aerobic fitness at 12 weeks (end of intervention)
  Aerobic fitness (ml/kg/min) will be measured by maximal cardiopulmonary exercise test

SECONDARY OUTCOMES:
Change in physical activity levels | Change from baseline in physical activity at 12 weeks (end of intervention)
  Physical activity (minutes per week) will be measured by accelerometry
Change in hand grip strength | Change from baseline in hand grip strength at 12 weeks (end of intervention)
  Hand grip strength (kg) will be measured by as an estimate of overall body strength
Change in body Composition | Change from baseline in body composition at 12 weeks (end of intervention)
  Segmental body composition will be measured by bioelectrical impedence analysis. Sarcopenia will be assessment by PET-CT
Change in Dietary Intake | Change from baseline in dietary intake at 12 weeks (end of intervention)
  Food frequency questionnaire
Change in inflammatory status | Change from baseline in inflammatory status at 12 weeks (end of intervention)
  Blood samples will be analysed for inflammatory cytokines (TNF-alpha and interleukin (IL)-6 as measured by multi-plex assays
Change in energy metabolism | Change from baseline in energy metabolism at 12 weeks (end of intervention)
  Blood samples will be analysed for measures of energy metabolism (citrate secretion and lactate secretion)
Change in quality of Life | Change from baseline in quality of life at 12 weeks (end of intervention)
  EORTC questionnaire will be used to measure QOL

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Hussey, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- St James's Hospital, Dublin, Ireland

REFERENCES:
- [Derived] Kennedy SA, Annett SL, Dunne MR, Boland F, O'Neill LM, Guinan EM, Doyle SL, Foley EK, Elliott JA, Murphy CF, Bennett AE, Carey M, Hillary D, Robson T, Reynolds JV, Hussey J, O'Sullivan J. Effect of the Rehabilitation Program, ReStOre, on Serum Biomarkers in a Randomized Control Trial of Esophagogastric Cancer Survivors. Front Oncol. 2021 Sep 15;11:669078. doi: 10.3389/fonc.2021.669078. eCollection 2021. PMID 34604026
- [Derived] O'Neill LM, Guinan E, Doyle SL, Bennett AE, Murphy C, Elliott JA, O'Sullivan J, Reynolds JV, Hussey J. The RESTORE Randomized Controlled Trial: Impact of a Multidisciplinary Rehabilitative Program on Cardiorespiratory Fitness in Esophagogastric cancer Survivorship. Ann Surg. 2018 Nov;268(5):747-755. doi: 10.1097/SLA.0000000000002895. PMID 30004915